CLINICAL TRIAL: NCT04431778
Title: Evaluation of the Efficacy and Tolerance of Low Doses of Ethosuximide in the Treatment of Peripheral Neuropathic Pain
Acronym: E-PENEPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC-IR 2019 DELAGE
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Neuropathic Pain
Keywords: Ethosuximide; T-type calcium channel; Neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Ethosuximide

STUDY DESIGN:
Intervention Model Description: Randomisation 1:1 placebo or ethosuximide
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Placebo and ethosuximide will be indistinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethosuximide (Experimental): Patients with chronic peripheral neuropathic pain
  Interventions: Drug: Ethosuximide
- Placebo (Placebo Comparator): Patients with chronic peripheral neuropathic pain
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ethosuximide — Taking the treatment (1 daily intake during the evening meal) according to increasing dosage:
  Step 1: 2.5 ml (125 mg) / day for 7 days Step 2: 5 ml (250 mg) / day for 7 days Step 3: 7.5 ml (375 mg) / day for 7 days Step 4 (final): 10 ml (500 mg) / day for the remainder of the study (12 weeks).
  Arms: Ethosuximide
Drug: Placebo — Taking the treatment (1 daily intake during the evening meal) according to increasing dosage:
  Step 1: 2.5 ml (125 mg) / day for 7 days Step 2: 5 ml (250 mg) / day for 7 days Step 3: 7.5 ml (375 mg) / day for 7 days Step 4 (final): 10 ml (500 mg) / day for the remainder of the study (12 weeks).
  Arms: Placebo

SUMMARY:
Evaluation of the efficacy and tolerance of low doses of ethosuximide in the treatment of peripheral neuropathic pain

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled therapeutic trial evaluating the efficacy and safety of low doses of ethosuximide in neuropathic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (under effective contraception: pill, implant, IUD, sterilization) aged 18 years or older, suffering from peripheral neuropathic pain (DN4 ≥ 4) for more than 3 months, of intensity ≥ 4 on a numerical scale from 0 to 10, and whose analgesic treatment has been stable for more than a month,
* Patients affiliated to the French Social Security system,
* Patients whose free and informed consent has been obtained.

Exclusion Criteria:

* Pregnancy (βHCG+ blood) or breastfeeding,
* Neuropathic pain due to spinal cord or brain injury, phantom limb pain or algohallucinosis,
* Fibromyalgia or algodystrophy,
* Chronic pain syndrome that the patient cannot distinguish and/or is more intense than peripheral neuropathic pain,
* Significant abnormalities in liver (transaminases > 3N, cholestasis) and renal (MDRD < 60 mL/min) tests,
* Ongoing comorbidities: cancer, neurodegenerative pathology
* Severe depressive disorder in progress (as determined by the clinician), history of suicide attempts or hospitalization for depression,
* Diabetic patients (contraindicated due to the high sugar concentration of ethosuximide, 3g / 5 ml),
* Patients who have previously received ethosuximide (epilepsy or clinical trial),
* Surgery planned throughout the entire trial,
* Medical and surgical history incompatible with the study,
* Dependence on alcohol and/or drugs (for compliance purposes),
* Known allergy to succinimides (ethosuximide, methsuximide, phensuximide),
* Psychotic disorders,
* Epileptic patients,
* Patients benefiting from a legal protection measure (curatorship, guardianship, deprived of liberty or subject to judicial safeguard).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain intensity | Day 0
  Variation in pain intensity (NRS, Numerical Rating Scale 0-10) averaged over the 7 days prior to the start of treatment (D0) and over the last 7 days of treatment (12 weeks).
Neuropathic pain intensity | Day 84
  Variation in pain intensity (NRS, Numerical Rating Scale 0-10) averaged over the 7 days prior to the start of treatment (D0) and over the last 7 days of treatment (12 weeks).

SECONDARY OUTCOMES:
Patient's Global Impression of Change (PGIC scale) | Day 0, Day 28, Day 56, Day 84
  Assessment of the patient's feelings about the effectiveness of the treatment.
Health related quality of life | Day 0, Day 28, Day 56, Day 84
  Assessment of the patient's quality of life with EQ-5D-3L questionnaire
Quantitative sensory testing (QST) | Day 0, Day 28, Day 56, Day 84
  Assessment of mechanical sensitivity using the von Frey test (static allodynia) and the brush test (dynamic allodynia).
adverse event | Throughout the study
  Assessment of the tolerability of the treatment by patients and clinicians

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - University Hospital Lyon sud - Pierre Bénite, Lyon, AURA
  - Uniervity hospital, Amiens, Amiens
  - Hospital of Annecy Genevois, Annecy
  - University hospital, clermont ferrand, Clermont-Ferrand
  - CIC, Hospital University, Clermont Ferrand, Clermont-Ferrand
  - University Hospital, Grenoble, Grenoble
  - CHu Limoges, Limoges
  - Hospital University, Lyon, Lyon
  - University Hospital, Saint Etienne, Saint-Etienne
  - Hospital of Valence, Valence
  - Hospital of Voiron, Voiron